CLINICAL TRIAL: NCT05298137
Title: Passive Leg Raise for Pediatric Peripheral IV Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jonathan Gamble, Executive Director of Research for the Department of Anesthesiology, College of Medicine, University of Saskatchewan, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Bio #3221
Record Dates: First submitted 2022-03-06; First posted 2022-03-28 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia; Children, Only
Keywords: Pediatrics; Anesthesiology; Cannula; Anesthesia, Intravenous; Catheterization

STUDY DESIGN:
Intervention Model Description: The investigators propose a prospective, parallel group, open-label randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV Cannulation Without Passive Leg Raise (No Intervention): Patients will be randomized to either the passive leg raise (PLR) group or standard care (control group). In both groups baseline measurements of a peripheral vein diameter using ultrasound will be undertaken at the level of the left antecubital fossa with and without a proximally placed venous tourniquet.
  Those in the control group will then have a peripheral IV (PIV) placed in the ipsilateral arm as the baseline measurements, the number of attempts to successful PIV placement will be recorded. A repeat diameter assessment of the previously assessed vein, number of PIV attempts, and time to successful IV cannulation (measured as the time from skin puncture to successful IV cannulation) will be recorded.
- IV Cannulation With Passive Leg Raise (Experimental): Patients will be randomized to either the passive leg raise (PLR) group or standard care (control group). In both groups baseline measurements of a peripheral vein diameter using ultrasound will be undertaken at the level of the left antecubital fossa with and without a proximally placed venous tourniquet.
  Those in the passive leg raise (PLR) group will have their legs elevated to 45 degrees until successful peripheral IV (PIV) placement. A repeat diameter assessment of the previously assessed vein, number of PIV attempts, and time to successful IV cannulation (measured as the time from skin puncture to successful IV cannulation) will be recorded.
  Interventions: Procedure: Passive Leg Raise

INTERVENTIONS:
Procedure: Passive Leg Raise — A passive leg raise (PLR) is defined as raising a patient's legs to a 45-degree angle at the hip while supine.
  Arms: IV Cannulation With Passive Leg Raise

SUMMARY:
The investigators hypothesize peripheral intravenous cannulation (insertion of tube into vein) will be facilitated (decreases the number of attempts) by a passive leg raise (raising the legs at the hip to 45 degree in a child laying on their back) in children.

DETAILED DESCRIPTION:
Establishing peripheral intravenous (PIV) access in the pediatric population is challenging even in the hands of skilled practitioners.

A passive leg raise (PLR), raising a patient's legs to a 45 degree angle while supine, auto-transfuses the blood volume within the patient's lower extremities into the central venous compartment. Increasing the blood volume in the central venous compartment may also increase the volume and caliber of upper extremity peripheral veins. It remains to be studied whether a PLR increases peripheral vein diameter and if this would facilitate the placement of PIVs in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3 months to 17 years.
* American Society of Anesthesiology (ASA) physical status 1-3 scheduled for elective surgical procedures under general anesthesia.

Exclusion Criteria:

* Children undergoing procedures who already have adequate IV access (ie pre-established central or peripheral access).
* Those greater than the age of 17, as this is the age limit for care at the Jim Pattison Children's Hospital.
* Those with any lower limb pathology that limits range of motion.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 234 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
The number of attempts to successful catheterization. | During the intraoperative procedure.
  The study's primary outcome (number of peripheral IV attempts) will be analyzed using a Chi-square test.

SECONDARY OUTCOMES:
The mean change in peripheral vein diameter following passive leg raise, assessed on ultrasonography. | During the intraoperative procedure.
  The change, if any, in peripheral vein diameter will be measured by comparing the diameter assessed by ultrasound at baseline and following leg raise. Results will be compared using the student's t test.
Time from skin puncture to the confirmation of a functioning peripheral line. | Measured intraoperatively, an expected estimated average of 2 minutes.
  Time to vein cannulation will be compared using the student's t test.
Provider perception of PLR on vein visualization. | Immediately following successful cannulation in the experimental group.
  Chi-square testing will be used to evaluate provider perception of passive leg raise on vein visualization and palpation.
Provider perception of PLR on vein palpation. | Immediately following successful cannulation in the experimental group.
  Chi-square testing will be used to evaluate provider perception of passive leg raise on vein visualization and palpation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J Gamble, MD, Principal Investigator — Department of Anesthesiology, University of Saskatchewan
Locations (1):
- Jim Pattison Children's Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate results will be presented in manuscript form but no individual participant data (IPD) will be shared.